CLINICAL TRIAL: NCT03236337
Title: Effectiveness of MOVI Interventions on Improving Adiposity, Cognition and Subclinical Atherosclerosis by Increasing Aerobic Cardiorespiratory Fitness: MOVI-daFit
Brief Title: Effectiveness of MOVI Interventions on Adiposity, Cognition and Subclinical Atherosclerosis: MOVI-daFit!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI16/01919
Record Dates: First submitted 2017-07-21; First posted 2017-08-01 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity; Obesity; Children; Cardiovascular; Cardiorespiratory Fitness
Keywords: Physical activity; Obesity; Children; Cognitive function; Academic achievement; Cardiorespiratory fitness; Adiposity; Cardiovascular fitness; Atherosclerosis; Aerobic capacity
MeSH Terms: conditions — Motor Activity; Obesity; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention
- MOVI intervention (Experimental): - MOVI-da Fit! is a high intensity interval training intervention that consists on: a) 4 h/week of a standardized recreative, non-competitive physical activity extracurricular program; and b) informative sessions to parents and teachers about how schoolchildren can became more active. It is aimed to enhance physical fitness, motor skills, physical activity time and active behaviours among 9-to-11 years old children.
  Interventions: Behavioral: MOVI intervention

INTERVENTIONS:
Behavioral: MOVI intervention — MOVI-da Fit! is a multidimensional intervention that consists on: a) 4h/week of a standardized recreative, non-competitive physical activity extracurricular program; and b) informative sessions to parents and teachers about how schoolchildren can became more active. It is aimed to enhance physical fitness, motor skills, physical activity time and active behaviours among 9-to-11 years old children.
  Other Names: MOVI-da Fit!
  Arms: MOVI intervention

SUMMARY:
Project which objective is to test the effectiveness of an extracurricular physical activity intervention based on high intensity interval training (MOVI-daFit!) on improving cardiorespiratory fitness (CRF), cardiometabolic risk, executive function, and academic performance.

DETAILED DESCRIPTION:
In the last decade, this research group has tested the effectiveness of three interventions following this model. The first one (MOVI) was carried out in peripuberal age children (4th and 5th year of primary education, 8-11 years) and showed a moderate effect in reducing the adiposity of schoolchildren with higher BMI, an improvement of the lipid profile, without significantly improving the global cardiometabolic risk because it did not produce a reduction in insulinemia.

The second edition (MOVI-2), carried out at schoolchildren of the same age range, increased the duration and intensity of the sessions, and was focused on the development of muscular strength in order to improve insulinemia levels. The intervention showed proved effectiveness; in addition, the data from this intervention showed a modest improvement in girls' aerobic capacity, but not in boys.

The last edition (MOVI-KIDS) was aimed at children aged 4 to 7 years to test the hypotheses that vigorous physical activity at early ages could produce lifelong cardio-metabolic benefits. Data submitted for publication in this study show that, as in the case of the IDEFICS study in children of similar age, the intervention was not effective in improving fitness.

This new edition (MOVI-daFit!) has been designed as controlled cluster-randomized trial including 10 schools from Cuenca province, Spain. Five schools will be randomized to intervention group (IG), in which the intervention MOVI-daFit! will be conducted for children in fourth and fifth school grades (9-11 years old). The other five schools will be allocated to the control group (CG).

During an academic year the 4th and 5th schoolchildren allocated to IG will be carry out, in out of school hours, four times by week, one hour sessions of a standardized recreative, non competitive, physical activity intervention based on games adapted to high intensity interval training methodology (MOVI-daFit!). In the CG regular physical activity will continue.

At the end of the school year the researchers will determine main outcome variables: changes in VO2max, body fat by bioimpedance, reactive hyperemia index, academic achievement, executive function, and biochemical analytic procedures including lipid profile, insulin, HbA1, C ultrasensitive reactive protein and BDNF.

The hypotheses of this new edition will be that the MOVI-daFit! based on high intensity interval training (HITT) adapted for the 4th and 5th schoolchildren, will:

1. Increase the aerobic capacity (VO2max).
2. Reduce the percentage of body fat in the GI versus the GC by 6%.
3. Improve executive function and academic performance.
4. Improve subclinical markers of atherosclerosis (endothelial function and carotid intima-media thickness).

ELIGIBILITY:
Inclusion criteria:

* Schools must have at least one full classrooms for both the 4th and 5th grade of primary school.
* The approval of boards of governors will be necessary.
* Children's parents or legal representatives will sign an informed consent to participate.
* Parents will be invited to collaborate by filling in questionnaires with regard to family leisure habits, sleeping, eating and getting around town.

Exclusion criteria:

* Severe Spanish language learning difficulties.
* Serious physical or mental disorders identified by parents or teachers that would impede participation in the programme's activities.
* Children diagnoses of chronic disorders, such as heart disease, diabetes or asthma, which in the opinion of their paediatricians would prevent their participation in the programme's activities (MOVI-daFit!).

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 570 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
VO2 max | One year
  It will be assessed by using 20-m shuttle run test, which is validated to measure maximal aerobic capacity in children from 5 years.

SECONDARY OUTCOMES:
BDNF blood determination | One year
  Biochemical determinations will be performed in order to determine Brain-derived neurotrophic factor. It is a protein that, in humans, is encoded by the BDNF gene. BDNF acts on certain neurons of the central nervous system and the peripheral nervous system, helping to support the survival of existing neurons, and encourage the growth and differentiation of new neurons and synapses. In the brain, it is active in the hippocampus, cortex, and basal forebrain-areas vital to learning, memory, and higher thinking.
Health-related quality of life | One year
  By using the KIDSCREEN-27 for children from 8 years.
Sleep behaviors and sleep problems by questionnaire | One year
  By using the Spanish version of the Children's Sleep Habits Questionnaire (CSHQ) completed by parents. Four questions will be added in order to ask about bedtime, waking up, getting up, and total number of hours of sleep.
Sleep quality by accelerometry | One year
  The latency, quantity, duration of sleep and the number of awakenings will also be measured by accelerometry in a subsample of 242 school children.
  Actigraphy (ACT) is a non-invasive method used to study sleep-wake patterns and circadian rhythms by assessing movement. The GENEActive (ActivInsights) monitor will be used, a wristwatch device that monitors activity levels for extended continuous periods.
Motor skills | One year
  By using the Movement Assessment Battery for Children 2 (M-ABC 2)
Physical activity | One year
  In a sub-sample of 242 randomly selected school children will be measured objectively by GENEActive (ActivInsights) accelerometers during seven consecutive days (including nights), with a fixed frequency of 85.7Hz to collect raw acceleration data measured in g for each axis of motion (x, y, z).
Body fat% | One year
  Body fat percentage measured by Bioimpedance analysis
Academic achievement | One year
  Children´s mean scores on mathematics and language will be considered
Arterial Stiffness | One year
  Carotid intima-media thickness measurement through Sonosite Micromax ultrasound (Sonosite Inc., Bothell, Washington, USA).
Pulse wave velocity | One year
  Pulse wave velocity measurement through SphymgoCor System (AtCor Medical Pty Ltd Head Office, West Ryde, Australia)
Subclinical atherosclerosis | One year
  Reactive Hyperemia index measurement through ENDO- PAT (Moerland et al. Int J Vasc Med, 2012; 17; 682-86)
Executive function | One year
  Executive function will be measured by standardized tests using the NIH toolbox
Glucose profile | One year
  Glucose (mg/dl) level will be determined by using a system Cobas 8000 of Roche Diagnostics
Lipid profile | One year
  Apolipoproteins (mg/dl) level will be determined by using a system Cobas 8000 of Roche Diagnostics.
Insulin profile | One year
  Insulin (µU/L) level will be determined by using the Architect platform of Abbott ®
Ultrasensitive protein profile | One year
  C-reactive protein ultrasensitive (mg/l) level will be determined by using a system Cobas 8000 of Roche Diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Martínez-Vizcaíno, PhD, MD, Principal Investigator — Social and Health Care Research Center, University of Castilla-La Mancha
Locations (2):
- Spain (2):
  - Health and Social Research Centre, University of Castilla-La Mancha, Cuenca
  - Mairena Sánchez-López, Cuenca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Visier-Alfonso ME, Jimenez-Lopez E, Rodriguez-Gutierrez E, Mesas AE, Nunez de Arenas-Arroyo S, Diaz-Goni V, Alvarez-Bueno C, Martinez-Vizcaino V. Internal Consistency and Validity of a Short Spanish Version (10-Items) of the Center for Epidemiological Studies Depression Scale for Children and Adolescents (CES-DC). Depress Anxiety. 2024 Sep 25;2024:5409747. doi: 10.1155/2024/5409747. eCollection 2024. PMID 40226705
- [Derived] Pozuelo-Carrascosa DP, Martinez-Vizcaino V, Torres-Costoso A, Martinez MS, Rodriguez-Gutierrez E, Garrido-Miguel M. "Fat but Fit" Paradox and Cardiometabolic Risk in Children: The Role of Physical Activity. Child Obes. 2023 Jun;19(4):282-291. doi: 10.1089/chi.2022.0073. Epub 2022 Jul 26. PMID 35881859
- [Derived] Martinez-Vizcaino V, Garrido-Miguel M, Redondo-Tebar A, Notario-Pacheco B, Rodriguez-Martin B, Sanchez-Lopez M. The "Fat but Fit" Paradigm from a Children's Health-Related Quality of Life Perspective. Child Obes. 2021 Oct;17(7):449-456. doi: 10.1089/chi.2021.0041. Epub 2021 May 18. PMID 34009010